CLINICAL TRIAL: NCT06252701
Title: Assessing the Feasibility and Acceptability of the Reduction of Ultra-processed Foods From the Diets of a Subset of Patients With Depression - A Pilot Open Label Crossover Trial.
Brief Title: Diet and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-39884
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Depression; Major Depressive Disorder; Weight Gain; Obesity; Metabolic Syndrome
Keywords: Ultra-processed Food; Depression; Diet
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Weight Gain; Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: A pilot open label crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention diet then regular diet (Experimental): 4 weeks eating a diet low in ultra-processed foods in diet followed by 4 weeks of eating the participant's regular diet.
  Interventions: Behavioral: Reduction of Ultra-processed foods
- Regular diet then intervention diet (Experimental): 4 weeks of eating the participant's regular diet followed by 4 weeks of eating a diet low in ultra-processed foods.
  Interventions: Behavioral: Reduction of Ultra-processed foods

INTERVENTIONS:
Behavioral: Reduction of Ultra-processed foods — Reduction of Ultra-processed foods for four weeks.

SUMMARY:
This study is a pilot open label crossover trial to assess the feasibility and acceptability of reducing ultra- processed foods (UPF) in a personalized manner from the diets of patients with major depressive disorder who eat a large percentage of UPF.

DETAILED DESCRIPTION:
There is a need for additional treatment or augmentation strategies for people who have depression. Epidemiological and observational studies show that an increased consumption of ultra-processed food (UPF) is associated with an increased risk of developing depression. This study will test the hypothesis that that reducing UPF intake from the diets of patients with major depressive disorder who eat a large percentage of UPF is a feasible and acceptable intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year olds (inclusive), all race/ethnic groups
* Willing to not change psychotropic medication or psychotherapy regimen during the study
* Willing and able to come to UCSF for in person visits two times
* Ability to speak and read English and answer participant surveys

Exclusion Criteria:

* Psychiatric hospitalization in past 3 months
* Active suicidal ideation with intent and plan or scoring a 3 or higher on the Columbia suicide severity rating scale (C-SSRS)
* In a current severe mood state when entering the study that would prohibit compliance with study visits or dietary program
* Known GI abnormalities or known GI medical problems (diarrhea, chronic intestinal disease, toxic megacolon, ileum) or known swallowing or chewing disorders or issues
* Anticipating or planning any major changes in physical activity or sleep during the study
* Pregnant or planning to be pregnant during the study
* Breastfeeding or planning to breastfeed during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | 4 weeks and 9 weeks
  Percent of enrolled of participants who have reduced their ultra-processed food intake
Acceptability of the intervention | 4 weeks and 9 weeks
  Participant mean rating of ease of completing the intervention. The score range is 0-10 with 0 being very difficult to 10 being very easy.

CONTACTS AND LOCATIONS:
Overall Officials: D. Nyasha Chagwedera, MD, PhD, Principal Investigator — University of California, San Francisco; Andrew Krystal, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez-Donoso C, Sanchez-Villegas A, Martinez-Gonzalez MA, Gea A, Mendonca RD, Lahortiga-Ramos F, Bes-Rastrollo M. Ultra-processed food consumption and the incidence of depression in a Mediterranean cohort: the SUN Project. Eur J Nutr. 2020 Apr;59(3):1093-1103. doi: 10.1007/s00394-019-01970-1. Epub 2019 May 4. PMID 31055621
- [Background] Adjibade M, Julia C, Alles B, Touvier M, Lemogne C, Srour B, Hercberg S, Galan P, Assmann KE, Kesse-Guyot E. Prospective association between ultra-processed food consumption and incident depressive symptoms in the French NutriNet-Sante cohort. BMC Med. 2019 Apr 15;17(1):78. doi: 10.1186/s12916-019-1312-y. PMID 30982472
- [Background] Lane MM, Gamage E, Travica N, Dissanayaka T, Ashtree DN, Gauci S, Lotfaliany M, O'Neil A, Jacka FN, Marx W. Ultra-Processed Food Consumption and Mental Health: A Systematic Review and Meta-Analysis of Observational Studies. Nutrients. 2022 Jun 21;14(13):2568. doi: 10.3390/nu14132568. PMID 35807749
- [Background] Hecht EM, Rabil A, Martinez Steele E, Abrams GA, Ware D, Landy DC, Hennekens CH. Cross-sectional examination of ultra-processed food consumption and adverse mental health symptoms. Public Health Nutr. 2022 Nov;25(11):3225-3234. doi: 10.1017/S1368980022001586. Epub 2022 Jul 28. PMID 35899785
- [Background] Zheng L, Sun J, Yu X, Zhang D. Ultra-Processed Food Is Positively Associated With Depressive Symptoms Among United States Adults. Front Nutr. 2020 Dec 15;7:600449. doi: 10.3389/fnut.2020.600449. eCollection 2020. PMID 33385006
- [Background] Pagliai G, Dinu M, Madarena MP, Bonaccio M, Iacoviello L, Sofi F. Consumption of ultra-processed foods and health status: a systematic review and meta-analysis. Br J Nutr. 2021 Feb 14;125(3):308-318. doi: 10.1017/S0007114520002688. Epub 2020 Aug 14. PMID 32792031
- [Background] Mazloomi SN, Talebi S, Mehrabani S, Bagheri R, Ghavami A, Zarpoosh M, Mohammadi H, Wong A, Nordvall M, Kermani MAH, Moradi S. The association of ultra-processed food consumption with adult mental health disorders: a systematic review and dose-response meta-analysis of 260,385 participants. Nutr Neurosci. 2023 Oct;26(10):913-931. doi: 10.1080/1028415X.2022.2110188. Epub 2022 Sep 12. PMID 36094005